CLINICAL TRIAL: NCT01473940
Title: Ipilimumab and Gemcitabine for Advanced Pancreas Cancer: A Phase Ib Study
Brief Title: Ipilimumab and Gemcitabine Hydrochloride in Treating Patients With Stage III-IV or Recurrent Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Principal Investigator, Mary Mulcahy, Mary Mulcahy, MD, Northwestern University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 10I02; NCI-2011-03135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00045323 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-10-19; First posted 2011-11-17 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody, chemotherapy) (Experimental): INDUCTION: Patients receive ipilimumab IV over 90 minutes in weeks 1, 4, 7, and 10 and gemcitabine hydrochloride IV over 30 minutes in weeks 1-7 and 9-11.
  MAINTENANCE: Beginning in week 22, patients receive ipilimumab IV over 90 minutes once every 12 weeks and gemcitabine hydrochloride IV over 30 minutes once weekly for 3 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  Interventions: Biological: ipilimumab; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab when given together with gemcitabine hydrochloride in treating patients with stage III-IV or recurrent pancreatic cancer that cannot be removed by surgery. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or tumor-killing substances to them. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to kill tumor cells or stop them from growing. Giving monoclonal antibody therapy together with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of ipilimumab.

INDUCTION: Patients receive ipilimumab intravenously (IV) over 90 minutes in weeks 1, 4, 7, and 10, and gemcitabine hydrochloride IV over 30 minutes in weeks 1-7 and 9-11.

MAINTENANCE: Beginning in week 22, patients receive ipilimumab IV over 90 minutes once every 12 weeks and gemcitabine hydrochloride IV over 30 minutes once weekly for 3 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.

After completion of study treatment, patients are followed up monthly for 6 months and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Histologic or cytologic diagnosis of pancreas adenocarcinoma advanced or recurrent (stage III or IV) that is unresectable; histologic or cytologic pathology from any prior surgery is sufficient for diagnosis
* Must have measurable disease by modified WHO criteria
* White blood cells (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100 x 10^3/uL
* Hemoglobin >= 9 g/dL (>= 80 g/L; may be transfused)
* Creatinine =< 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Bilirubin =< 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-1
* Prior systemic therapy for advanced pancreas cancer with gemcitabine is prohibited; prior gemcitabine with radiotherapy for localized pancreas cancer is allowed provided disease is present outside of the radiated field; prior gemcitabine as adjuvant therapy to surgical resection is allowed provided 3 months or greater has elapsed between the last dose of gemcitabine and the detection of recurrent disease
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal; post-menopause is defined as: amenorrhea >= 12 consecutive months without another cause, or for women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL; women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotrophin [HCG]) within 72 hours before the start of ipilimumab
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized
* Patients on stable anticoagulation are eligible for enrollment; for patients on warfarin, prothrombin time (PT)/international normalized ratio (INR) should be monitored every 2 weeks during induction therapy, monthly thereafter, or more frequent as clinically indicated

Exclusion Criteria:

* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis)
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with ipilimumab or prior tumor necrosis factor receptor superfamily, member 9 (CD137) agonist or cytotoxic T-lymphocyte-associated protein 4 (CTLA4) inhibitor or agonist
* Concomitant therapy with any of the following: interleukin (IL)2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids
* WOCBP who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness
* Patients with symptoms of partial or complete bowel obstruction and recent (within 6 month) history of fistula, intra-abdominal abscess or bowel perforation
* Patients with a history or evidence of central nervous system (CNS) disease, including brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Patients currently receiving radiation therapy or those having received radiation within 4 weeks of study entry
* Patients with any known active infection or known history of tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2014-10-16 (Actual); Study Completion 2018-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened at our site April 3, 2012 with the first patient being enrolled and starting treatment on June 11, 2012. The study was designed to with 4 dose escalation cohorts to determine maximum tolerated dose (MTD) and then an expansion cohort at the MTD. The study closed March 23, 2016 with a total of 21 patients treated on the study.
Groups:
- Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg; Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg; Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg; Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg: INDUCTION: Patients receive ipilimumab IV over 90 minutes in weeks 1, 4, 7, and 10 and gemcitabine hydrochloride IV over 30 minutes in weeks 1-7 and 9-11.
  MAINTENANCE: Beginning in week 12, patients receive ipilimumab IV over 90 minutes once every 12 weeks and gemcitabine hydrochloride IV over 30 minutes once weekly for 3 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  Ipilimumab: Given IV
  Gemcitabine hydrochloride: Given IV
Period: Induction Therapy
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
Started | 3 | 4 | 6 | 8
Started Treatment | 3 | 4 | 6 | 8
Completed Induction- 12 Weeks | 3 | 3 | 4 | 7
Completed | 3 | 3 | 4 | 7
Not Completed | 0 | 1 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Progressive Disease | 0 | 1 | 1 | 0
Period: Maintenance Therapy
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
Started | 3 | 3 | 4 | 7
Evaluated for Response | 3 | 3 | 4 | 7
Went on to Start Maintenance Therapy | 2 | 1 | 3 | 3
Completed | 2 | 1 | 3 | 3
Not Completed | 1 | 2 | 1 | 4
Not completed — Progressive Disease | 1 | 2 | 1 | 4
Period: Follow-up Until Death
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
Started (All patients that receive at least one dose of study treatment go into the follow up phase.) | 3 | 4 | 5 | 7
Completed | 3 | 4 | 5 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 2 | 9
  >=65 years | 2 | 1 | 3 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 4 | 13
  Male | 1 | 1 | 2 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 6 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 5 | 6 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 6 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) Seen in Patients With Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination in Order to Define the Maximum Tolerated Dose (MTD)
Description: Dose limiting toxicity (DLT) will be monitored by calculating the Bayesian predictive probability of a DLT given the data to date. All toxicities will be summarized in a descriptive manner as to type, frequency, attribution and timing by dose level. Safety will be evaluated for all treated patients using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 where grading is as follows:
  Mild (grade 1) Moderate (grade 2) Severe (grade 3) Life-threatening (grade 4) Fatal (grade 5)
  In general a DLT will be defined as any any of the following drug-related toxicities:
  Febrile neutropenia with grade 3/4 neutropenia Asymptomatic grade 4 neutropenia more than 7 days Grade 3 thrombocytopenia with grade 3-4 hemorrhage or grade 4 thrombocytopenia Non-hematologic toxicity grade 3 or 4 (with some protocol specified exceptions)
  DLTs will be used to determine the MTD for the expansion cohort of the study.
  *AST = Aspartate transamina
Time Frame: During the 12 weeks of Induction Therapy
Measure: Number; unit: DLTs
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg
Number analyzed (Participants) | 3 | 4 | 6
DLTs
  Number of DLTS seen in cohort | 0 | 0 | 2
  Number of AST increase DLTs seen in cohort | 0 | 0 | 1
  Number of diarrhea DLTs seen in cohort | 0 | 0 | 1
Statistical Analysis 1: Comparison: Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg vs Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg vs Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg; A 3 + 3 enrollment design was adopted to monitor safety and determine the MTD based on DLTs obsesved. The MTD is the highest dose at which 0 of 3 or 1 of 6 DLTs are detected. The MTD is exceeded if 2 of 3 or 2 of 6 DLTs are detected. There will be no dose escalation within a cohort; Test type: Other; P-Value not used; The number of DLTs seen at each cohort were used to determine the MTD for the expansion cohort. The MTD was determined to be Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg

2. Secondary Outcome: Response Rate Using Immune-related Response Criteria (irRC) in Patients With Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination
Description: Response will be assessed using CT of MRI scans immune-related response criteria (irRC). The sum of all the products of diameters (SPD) at tumor assessment using the irRC for progressive disease incorporates the contribution of new measurable lesions. Each net percentage change in tumor burden per assessment using irRC accounts for the size and growth kinetics of both old and new lesions as they appear.
  irComplete Response (irCR)-Complete disappearance of all index lesions. irPartial Response (irPR)-Decrease of 50% or greater in the sum of products of the two largest perpendicular diameters of all index and all new measurable lesions (i.e., percentage change in tumor burden) irStable Disease (irSD)-does not meet criteria for irCR or ir PR, in the absence of progressive disease.
  irProgressive Disease (irPD)-At least 25% increase in the percentage change in tumor burden (i.e., taking sum of all the products of all the index lesions and any new lesions) when compared to SPD at nadir.
Time Frame: Every 12 weeks during treatment with a 12 week induction and then 28 day maintenance cycles. Range of cycles completed (including induction cycle) 0-10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 6 | 8
Participants
  irCR | 0 | 0 | 0 | 0
  irPR | 0 | 1 | 1 | 1
  irSD | 2 | 0 | 3 | 2
  irPD | 1 | 3 | 1 | 3
  NE - Death | 0 | 0 | 1 | 2

3. Secondary Outcome: Time to Progression Patients With Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination Who Progress While on Treatment
Description: Time to Progression will be defined as the time from treatment initiation until the first documentation of progression as calculated by irRC in patients who show progression. Progression will be defined as at least a 25% increase percentage change in tumor burden (i.e., taking the sum of all the products of all index lesions and any new lesions) when compared to sum of all the products of diameters (SPD) at nadir.
Time Frame: as for outcome 2
Population: PFS was considered to be a more meaningful outcome measure to report on. This outcome measure was so similar that it was considered duplicate information and data was not collected and analyzed specifically for this outcome measure.
Groups:
- Cohort 2/Expansion Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg; Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg: INDUCTION: Patients receive ipilimumab IV over 90 minutes in weeks 1, 4, 7, and 10 and gemcitabine hydrochloride IV over 30 minutes in weeks 1-7 and 9-11.
  MAINTENANCE: Beginning in week 12, patients receive ipilimumab IV over 90 minutes once every 12 weeks and gemcitabine hydrochloride IV over 30 minutes once weekly for 3 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  Ipilimumab: Given IV
  Gemcitabine hydrochloride: Given IV
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2/Expansion Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS) in Patients With Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination
Description: Median Progression Free Survival (mPFS) was estimated using a Kaplan-Meier curve with 0 censored patients. PFS is defined from the time of treatment initiation until the first documentation of progressive disease. Any patient without the event at the time of analysis will be censored from the last documented contact.
Time Frame: as for outcome 2
Population: Cohort 2 and expansion cohorts are combined for this outcome measure as they were both at the MTD doses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2/Expansion Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg
Number analyzed (Participants) | 3 | 12 | 6
months | 3.3859 [2.5970 to 8.0868] | 2.5312 [0.7890 to 4.8323] | 3.8626 [0.7561 to 22.4195]

5. Secondary Outcome: Overall Survival (OS) in Patients With Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination
Description: Overall Survival (OS) was estimated using a kaplan-meier curve with 0 patients censored. OS is defined from the time of treatment initiation until the time of death from any cause. Any patient without the event at the time of analysis will be censored from the last documented contact.
Time Frame: as for outcome 2
Population: Cohort 2 and expansion cohorts are combined for this outcome measure as they were both at the MTD doses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2/Expansion Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg
Number analyzed (Participants) | 3 | 12 | 8
months | 5.3254 [5.0953 to 9.5661] | 5.7199 [1.6108 to 22.8139] | 8.9908 [0.7561 to 30.0460]

6. Secondary Outcome: Recovery of Tumor Immune Surveillance: T-cell Response to Defined Pancreatic Cancer Tumor Antigens
Description: Optional blood draws to analyze the inflammatory T cell function before, during and after treatment.
Time Frame: Prior to ipilimumab infusion at weeks 1, 4, 7, and 10, and then every 12 weeks starting at week 13 where range of cycles including induction cycle was 0-10 (Induction cycle = 12 weeks, maintenance cycle = 28 days)
Population: Due to this being optional, insufficient samples were obtained and no data or analysis of blood was completed.
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Post Hoc Outcome: Duration of Response in Patients Pancreas Adenocarcinoma Treated With Ipilimumab and Gemcitabine Combination
Description: Duration of response is shown below for patients who showed a response as defined by immune-related response criteria (irCR) as either of the following:
  irComplete Response (irCR)-Complete disappearance of all index lesions or irPartial Response (irPR)-Decrease of 50% or greater in the sum of products of the two largest perpendicular diameters of all index and all new measurable lesions (i.e., percentage change in tumor burden)
  Duration of response is defined as the time from first documentation of response to first documentation of progression, with progression defined as:
  irProgressive Disease (irPD)-At least 25% increase in the percentage change in tumor burden (i.e., taking sum of all the products of all the index lesions and any new lesions) when compared to the sum of all the product diameters (SPD) at nadir.
Time Frame: From the time of response and every 12 weeks during treatment with a 12 week induction and then 28 day maintenance cycles. Range of cycles completed (including induction cycle) 0-10
Population: Only patients with a response are shown here.
Measure: Number; unit: months
Groups:
- Cohort 2 Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg; Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg; Expansion - Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg: INDUCTION: Patients receive ipilimumab IV over 90 minutes in weeks 1, 4, 7, and 10 and gemcitabine hydrochloride IV over 30 minutes in weeks 1-7 and 9-11.
  MAINTENANCE: Beginning in week 12, patients receive ipilimumab IV over 90 minutes once every 12 weeks and gemcitabine hydrochloride IV over 30 minutes once weekly for 3 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.
  Ipilimumab: Given IV
  Gemcitabine hydrochloride: Given IV
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion - Gemcitabine-1,000mg/m2+Ipilimumab-3mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 1
months |  | 8.5 | 19.8 | 11

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of treatment initiation until treatment discontinuation for any reason. Treatment was considered to be one induction cycle of 12 weeks followed by 28 day maintenance cycles with the range of cycles completed by any patients 0-10 (including the induction cycle)
Arm/Group | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 8/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 4/6 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg (N=3) | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg (N=4) | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg (N=6) | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg (N=8)
Duodenal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter-related Infection (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Patient also with vomiting, hypokalemia and dehydration during this event
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 — Patient also with hypotension and fever during this event
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 (2) | 0 — Patient also with Abdominal pain during this event
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Patient also with portal hypertension at the time of the event
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Patient also with diarrhea at the time of the event
Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0
Sepsis resulting in death (Infections and infestations) | 0 | 0 | 1 | 0 — the patient was also with hypertension at the time of the event
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — This lead to a hematoma
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Patient also with vomiting and abdominal pain at the time of this event
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Patient also with vomiting at the time of the event
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 — Patient also with dehydration, hypotension, ascites and pleural effusion and died due to this SAE.
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Patient also with fever during this event.
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Facial Muscle Weakness (Nervous system disorders) | 0 | 0 | 0 | 1
Death due to disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Patient also with Abdominal pain during the event
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 — patient also with headache and tinnitus during the event
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Gemcitabine - 750 mg/m2, Ipilimumab 3 mg/kg (N=3) | Cohort 2 Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg (N=4) | Cohort 3 Gemcitabine -1,000 mg/m2, Ipilimumab 6 mg/kg (N=6) | Expansion Cohort Gemcitabine - 1,000 mg/m2, Ipilimumab 3 mg/kg (N=8)
Anemia (Blood and lymphatic system disorders) | 2 | 4 | 6 | 7
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 2 | 3 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear feels full (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Blurred Vision (Eye disorders) | 0 | 0 | 1 | 0
Watery Eyes (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 3 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 6 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 4 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 6 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Chills (General disorders) | 0 | 2 | 1 | 2
Edema in Limbs (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 2 | 6 | 6
Fever (General disorders) | 2 | 2 | 1 | 4
Flu-like Symptoms (General disorders) | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Papulpustular Rash (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 3 | 4 | 2
Alkaline Phosphatase Increased (Investigations) | 1 | 2 | 5 | 6
Aspartate Aminotransferase Increased (Investigations) | 2 | 3 | 6 | 6
Blood Bilirubin Increased (Investigations) | 1 | 2 | 3 | 2
Cardiac Troponin 1 Increased (Investigations) | 0 | 0 | 1 | 0
Creatinine Increased (Investigations) | 0 | 1 | 3 | 2
INR Increased (Investigations) | 1 | 1 | 3 | 0
Hyperlipidemia (Investigations) | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 3 | 4 | 5 | 4
Neutrophil Count Decreased (Investigations) | 2 | 2 | 5 | 3
Platelet Count Decreased (Investigations) | 2 | 4 | 6 | 5
Serum Amylase Increased (Investigations) | 1 | 0 | 0 | 0
Weight Gain (Investigations) | 0 | 1 | 0 | 0
Weight Loss (Investigations) | 2 | 2 | 2 | 1
White Blood Cell Decreased (Investigations) | 2 | 3 | 5 | 3
Anorexia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 6 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4 | 5 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4 | 4 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 1 | 0
Headaches (Nervous system disorders) | 0 | 1 | 1 | 3
Movements Involuntary (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Radiculitis (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomina (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hemaruria (Renal and urinary disorders) | 1 | 1 | 0 | 1
Uriary Discoloration (Renal and urinary disorders) | 1 | 1 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Tract Pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Maculo-papular Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 3 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hot Flashes (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tinnnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes